CLINICAL TRIAL: NCT04392219
Title: A Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study Designed to Evaluate the Safety, Tolerability, and Pharmacokinetics of EIDD-2801 Following Oral Administration to Healthy Volunteers
Brief Title: COVID-19 First In Human Study to Evaluate Safety, Tolerability, and Pharmacokinetics of EIDD-2801 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ridgeback Biotherapeutics, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EIDD-2801-1001; 2020-001407-17 (EudraCT Number)
Record Dates: First submitted 2020-04-29; First posted 2020-05-18 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus
Keywords: Coronavirus; EIDD-2801; ribonucleoside
MeSH Terms: conditions — Coronavirus Infections | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EIDD-2801 (Experimental): EIDD-2801: Part 1: Participants were randomized to receive 50 to 1600 mg EIDD-2801 powder-in bottle (fasted); Part 2: Participants were randomized to receive two single 200 mg doses (fed or fasted); Part 3: Participants were randomized to receive twice daily doses of EIDD-2801 in an open-label manner.
  Interventions: Drug: EIDD-2801
- Placebo (Placebo Comparator): Placebo: Part 1: Participants were randomized to receive placebo (fasted); Part 3: Participants were randomized to receive placebo (fasted).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EIDD-2801 — Part 1:
  Participants will be randomized to receive a single oral dose of EIDD-2801 or Placebo.
  Part 2:
  Two single oral doses of EIDD-2801 will be administered to participants, in an open-label manner.
  Part 3:
  Participants will be randomized to receive twice daily dosing either EIDD-2801 or Placebo.
  Other Names: Molnupiravir
  Arms: EIDD-2801
Drug: Placebo — Part 1:
  Participants will be randomized to receive a single oral dose of EIDD-2801 or Placebo.
  Part 3:
  Participants will be randomized to receive twice daily dosing either EIDD-2801 or Placebo.
  Arms: Placebo

SUMMARY:
This is a First In Human study designed to assess the safety, tolerability and pharmacokinetics of EIDD-2801 in healthy human volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, First-in-Human study designed to evaluate the safety, tolerability, and pharmacokinetics of EIDD-2801 following oral administration to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 60, inclusive.
* Female participants must be of non-childbearing potential.
* Male participants must agree to the use of effective contraception for study duration
* Is in generally good health as determined by medical history, physical examinations (PEs) (at Screening and/or Check-in), vital signs, and other screening procedures.
* Has a body mass index (BMI) of 18 to 30 kg/m^2.

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or breastfeeding.
* Has a clinically relevant acute or chronic medical condition or disease of the cardiovascular, gastrointestinal (GI), hepatic, renal, endocrine, pulmonary, neurologic, or dermatologic systems as determined by the principal investigator (PI) (or designee).
* Has any current or historical disease or disorder of the hematological system or significant liver disease or family history of bleeding/platelet disorders.
* Has a history of cancer (other than basal cell or squamous cell cancer of the skin), rheumatologic disease or blood dyscrasias.
* Has a history of gastrointestinal (GI) surgery or other condition that may interfere with absorption of study drug, in the opinion of the principal investigator (PI) (or designee).
* Has a history of febrile illness within the 14 days prior to the first dose of study drug.
* Has a positive alcohol or drug screen at Screening or the Day -1 visit or has a history of alcohol or drug abuse within the past 5 years.
* Currently uses tobacco, nicotine or tobacco products or e-cigarettes, or stopped using tobacco products within the past 3 months
* Has a total white cell count or absolute lymphocyte count outside the normal range, or hemoglobin or platelet levels below the lower limit of normal, at Screening or Day -1.
* Has values above the upper limit of normal for the following laboratory analytes: alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT), alkaline phosphatase (serum), aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), at Screening or Day -1.
* Positive test result for human immunodeficiency virus (HIV), hepatitis b virus (HBV), or hepatitis c virus (HCV).
* Has an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
* Has any of the following:

  * QT interval corrected for heart rate (using Fridericia's formula) (QTcF) >450 ms confirmed by repeat measurement
  * QRS duration >110 ms confirmed by repeat measurement
  * PR interval >220 ms confirmed by repeat measurements
  * findings which would make QTc measurements difficult or QTc data uninterpretable
  * history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
* Except as noted, has used prescription drugs (other than hormone replacement therapy) within 14 days prior to the first dose of study drug unless, in the opinion of the PI (or designee), the drug will not interfere with study assessments.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 3 months prior to the first dose of study drug and agrees not to receive another experimental agent during the duration of this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, Principal Investigator — Covance Clinical Research Unit Limited
Locations (1):
- Covance Leeds Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The same 10 participants started and completed the Part 200 mg EIDD-2801 (Fasted) and Part 200 mg EIDD-2801 (Fed) arms.
Groups:
- Part 1 - Placebo: Participants were randomized to receive a single oral dose of Placebo (fasted).
- Part 1 - 50 mg EIDD-2801: Participants were randomized to receive 50 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 100 mg EIDD-2801: Participants were randomized to receive 100 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 200 mg EIDD-2801: Participants were randomized to receive 200 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 400 mg EIDD-2801: Participants were randomized to receive 400 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 600 mg EIDD-2801: Participants were randomized to receive 600 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 800 mg EIDD-2801: Participants were randomized to receive 800 mg EIDD-2801 powder-in-bottle (fasted).
- Part 1 - 1200 mg EIDD-2801: Participants were randomized to receive 1200 mg EIDD-2801 capsule (fasted).
- Part 1 - 1600 mg EIDD-2801: Participants were randomized to receive 1600 mg EIDD-2801 capsule (fasted).
- Part 2 - 200 mg EIDD-2801 (Fasted/Fed): Participants were randomized to receive two single 200 mg oral doses of EIDD-2801 in an open-label manner (fasted/fed).
- Part 3 - Placebo: Participants were randomized to receive a twice daily dosing of Placebo capsules (fasted).
- Part 3 - 50 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 50-mg EIDD-2801 capsules (fasted).
- Part 3 - 100 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 100-mg EIDD-2801 capsules (fasted).
- Part 3 - 200 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 200-mg EIDD-2801 capsules (fasted).
- Part 3 - 300 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 300-mg EIDD-2801 capsules (fasted).
- Part 3 - 400 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 400-mg EIDD-2801 capsules (fasted).
- Part 3 - 600 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 600-mg EIDD-2801 capsules (fasted).
- Part 3 - 800 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 800-mg EIDD-2801 capsules (fasted).
Period: Overall Study
Arm/Group | Part 1 - Placebo | Part 1 - 50 mg EIDD-2801 | Part 1 - 100 mg EIDD-2801 | Part 1 - 200 mg EIDD-2801 | Part 1 - 400 mg EIDD-2801 | Part 1 - 600 mg EIDD-2801 | Part 1 - 800 mg EIDD-2801 | Part 1 - 1200 mg EIDD-2801 | Part 1 - 1600 mg EIDD-2801 | Part 2 - 200 mg EIDD-2801 (Fasted/Fed) | Part 3 - Placebo | Part 3 - 50 mg EIDD-2801 | Part 3 - 100 mg EIDD-2801 | Part 3 - 200 mg EIDD-2801 | Part 3 - 300 mg EIDD-2801 | Part 3 - 400 mg EIDD-2801 | Part 3 - 600 mg EIDD-2801 | Part 3 - 800 mg EIDD-2801
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Part 3 - Placebo: Participants were randomized to receive two daily dosing of Placebo capsules (fasted).
- Part 3 - 50 mg EIDD-2801: Participants were randomized to receive two daily dosing of 50 mg EIDD-2801 capsules (fasted).
- Part 3 - 100 mg EIDD-2801: Participants were randomized to receive two daily dosing of 100 mg EIDD-2801 capsules (fasted).
- Part 3 - 200 mg EIDD-2801: Participants were randomized to receive two daily dosing of 200 mg EIDD-2801 capsules (fasted).
- Part 3 - 300 mg EIDD-2801: Participants were randomized to receive two daily dosing of 300 mg EIDD-2801 capsules (fasted).
- Part 3 - 400 mg EIDD-2801: Participants were randomized to receive two daily dosing of 400 mg EIDD-2801 capsules (fasted).
- Part 3 - 600 mg EIDD-2801: Participants were randomized to receive two daily dosing of 600 mg EIDD-2801 capsules (fasted).
- Part 3 - 800 mg EIDD-2801: Participants were randomized to receive two daily dosing of 800 mg EIDD-2801 capsules (fasted).
- Total: Total of all reporting groups
Arm/Group | Part 1 - Placebo | Part 1 - 50 mg EIDD-2801 | Part 1 - 100 mg EIDD-2801 | Part 1 - 200 mg EIDD-2801 | Part 1 - 400 mg EIDD-2801 | Part 1 - 600 mg EIDD-2801 | Part 1 - 800 mg EIDD-2801 | Part 1 - 1200 mg EIDD-2801 | Part 1 - 1600 mg EIDD-2801 | Part 2 - 200 mg EIDD-2801 (Fasted/Fed) | Part 3 - Placebo | Part 3 - 50 mg EIDD-2801 | Part 3 - 100 mg EIDD-2801 | Part 3 - 200 mg EIDD-2801 | Part 3 - 300 mg EIDD-2801 | Part 3 - 400 mg EIDD-2801 | Part 3 - 600 mg EIDD-2801 | Part 3 - 800 mg EIDD-2801 | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 130
Age, Continuous [Mean (Full Range); unit: years] | 39.4 [22 to 56] | 52.0 [34 to 57] | 41.2 [23 to 58] | 39.8 [26 to 60] | 42.0 [23 to 57] | 38.2 [21 to 57] | 39.5 [23 to 56] | 34.2 [24 to 56] | 30.8 [25 to 46] | 45.3 [30 to 60] | 37.5 [19 to 59] | 34.0 [23 to 56] | 45.5 [20 to 58] | 36.8 [22 to 60] | 36.2 [20 to 58] | 38.8 [20 to 60] | 30.8 [20 to 54] | 30.8 [20 to 58] | 38.7 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 21
  Male | 14 | 4 | 4 | 5 | 4 | 4 | 6 | 6 | 6 | 7 | 12 | 5 | 5 | 6 | 4 | 5 | 6 | 6 | 109
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  White | 16 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 5 | 9 | 13 | 6 | 6 | 5 | 5 | 6 | 6 | 5 | 122
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.80 (2.217) | 26.07 (2.649) | 23.50 (3.501) | 26.68 (2.320) | 24.48 (2.349) | 25.32 (1.847) | 26.45 (2.745) | 25.15 (1.623) | 23.37 (2.954) | 25.38 (2.185) | 24.79 (2.681) | 22.27 (3.371) | 24.97 (4.162) | 25.50 (3.117) | 24.48 (1.901) | 24.32 (2.866) | 24.50 (3.679) | 24.20 (2.504) | 24.81 (2.707)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events and Severity of Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events (TEAEs) and severity of TEAEs following a single dose of EIDD-2801 in Part 1
Time Frame: From screening through study completion, up to 15 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Placebo | Part 1 - 50 mg EIDD-2801 | Part 1 - 100 mg EIDD-2801 | Part 1 - 200 mg EIDD-2801 | Part 1 - 400 mg EIDD-2801 | Part 1 - 600 mg EIDD-2801 | Part 1 - 800 mg EIDD-2801 | Part 1 - 1200 mg EIDD-2801 | Part 1 - 1600 mg EIDD-2801
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  TEAEs (Overall) | 7 | 2 | 0 | 3 | 3 | 4 | 2 | 1 | 2
  Mild (Grade 1) | 7 | 2 | 0 | 3 | 3 | 4 | 2 | 1 | 2
  Moderate (Grade 2) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 3: Number of Participants With Treatment Emergent Adverse Events and Severity of Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events (TEAEs) and severity of TEAEs following multiple doses of EIDD-2801 in Part 3
Time Frame: From screening through study completion, up to 20 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Part 3 - Placebo: Participants were randomized to receive twice daily dosing of Placebo capsules (fasted).
- Part 3 - 50 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 50 mg EIDD-2801 capsules (fasted).
- Part 3 - 100 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 100 mg EIDD-2801 capsules (fasted).
- Part 3 - 200 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 200 mg EIDD-2801 capsules (fasted).
- Part 3 - 300 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 300 mg EIDD-2801 capsules (fasted).
- Part 3 - 400 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 400 mg EIDD-2801 capsules (fasted).
- Part 3 - 600 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 600 mg EIDD-2801 capsules (fasted).
- Part 3 - 800 mg EIDD-2801: Participants were randomized to receive twice daily dosing of 800 mg EIDD-2801 capsules (fasted).
Arm/Group | Part 3 - Placebo | Part 3 - 50 mg EIDD-2801 | Part 3 - 100 mg EIDD-2801 | Part 3 - 200 mg EIDD-2801 | Part 3 - 300 mg EIDD-2801 | Part 3 - 400 mg EIDD-2801 | Part 3 - 600 mg EIDD-2801 | Part 3 - 800 mg EIDD-2801
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  TEAEs (Overall) | 7 | 2 | 3 | 3 | 2 | 3 | 2 | 3
  Mild (Grade 1) | 7 | 2 | 3 | 3 | 2 | 3 | 2 | 3
  Moderate (Grade 2) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of the first study drug administration until the completion of the End of Study visit (Part 1: approximately 15 days, Part 2: approximately 30 days, and Part 3: approximately 20 days)
Description: Once each day while the participant was in the clinic and once during each out-patient visit, the principal investigator (or designee) inquired about the occurrence of adverse events.
  Open-ended questions may have been used to obtain this information.
Groups:
- Part 2 - 200 mg EIDD-2801 (Fasted): Participants were randomized to receive two single 200 mg oral doses of EIDD-2801 in an open-label manner (fasted).
- Part 2 - 200 mg EIDD-2801 (Fed): Participants were randomized to receive two single 200 mg oral doses of EIDD-2801 in an open-label manner (fed).
Arm/Group | Part 1 - Placebo | Part 1 - 50 mg EIDD-2801 | Part 1 - 100 mg EIDD-2801 | Part 1 - 200 mg EIDD-2801 | Part 1 - 400 mg EIDD-2801 | Part 1 - 600 mg EIDD-2801 | Part 1 - 800 mg EIDD-2801 | Part 1 - 1200 mg EIDD-2801 | Part 1 - 1600 mg EIDD-2801 | Part 2 - 200 mg EIDD-2801 (Fasted) | Part 2 - 200 mg EIDD-2801 (Fed) | Part 3 - Placebo | Part 3 - 50 mg EIDD-2801 | Part 3 - 100 mg EIDD-2801 | Part 3 - 200 mg EIDD-2801 | Part 3 - 300 mg EIDD-2801 | Part 3 - 400 mg EIDD-2801 | Part 3 - 600 mg EIDD-2801 | Part 3 - 800 mg EIDD-2801
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/10 | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/10 | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/16 | 2/6 | 0/6 | 3/6 | 3/6 | 4/6 | 2/6 | 1/6 | 2/6 | 2/10 | 1/10 | 7/14 | 2/6 | 3/6 | 3/6 | 2/6 | 3/6 | 2/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Placebo (N=16) | Part 1 - 50 mg EIDD-2801 (N=6) | Part 1 - 100 mg EIDD-2801 (N=6) | Part 1 - 200 mg EIDD-2801 (N=6) | Part 1 - 400 mg EIDD-2801 (N=6) | Part 1 - 600 mg EIDD-2801 (N=6) | Part 1 - 800 mg EIDD-2801 (N=6) | Part 1 - 1200 mg EIDD-2801 (N=6) | Part 1 - 1600 mg EIDD-2801 (N=6) | Part 2 - 200 mg EIDD-2801 (Fasted) (N=10) | Part 2 - 200 mg EIDD-2801 (Fed) (N=10) | Part 3 - Placebo (N=14) | Part 3 - 50 mg EIDD-2801 (N=6) | Part 3 - 100 mg EIDD-2801 (N=6) | Part 3 - 200 mg EIDD-2801 (N=6) | Part 3 - 300 mg EIDD-2801 (N=6) | Part 3 - 400 mg EIDD-2801 (N=6) | Part 3 - 600 mg EIDD-2801 (N=6) | Part 3 - 800 mg EIDD-2801 (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is required to obtain written consent from the Sponsor before anything relating to the study can be published.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT04392219/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04392219/SAP_001.pdf